CLINICAL TRIAL: NCT01902524
Title: Evaluation in Efficacy and Safety of Fentanyl-TTS (Durogesic® D-Trans) for Treatment of Chronic Pain
Brief Title: Efficacy and Safety Study of Fentanyl Transdermal Patch for Treatment of Chronic Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR002155; FEN-KOR-10 (Other: Janssen Korea, Ltd., Korea)
Record Dates: First submitted 2013-07-15; First posted 2013-07-18 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Chronic Pain
Keywords: Chronic Pain; Fentanyl-TTS; Fentanyl Patch; Transdermal; Non-cancer Pain
MeSH Terms: conditions — Chronic Pain | interventions — Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fentanyl-TTS (Experimental): Study drug administered in a form of one patch, either 21.0 cm2 or 10.5 cm2.
  Interventions: Drug: Fentanyl-TTS

INTERVENTIONS:
Drug: Fentanyl-TTS — All of the participants will receive the study drug at least once transdermally, administration dosage starts at 12.5 microgram/hour.
  Other Names: fentanyl

SUMMARY:
The purpose of this study is to confirm effectiveness and safety of fentanyl transdermal patch Durogesic® D-Trans for treatment of chronic pain in participants with chronic non-cancer pain.

DETAILED DESCRIPTION:
This trial is a Phase 4, prospective, open-label (meaning that both the research physician and study participants will know which medication is being administered) study of fentanyl transdermal patch-type system (TTS) Durogesic® D-Trans in patients with non-cancer pain. The patch is designed to systematically release the adsorbed fentanyl percutaneously, in a constant rate for three days (72 hours). The study will be conducted for 12 weeks. The efficacy and safety will be evaluated at week 1, week 4, week 8 and week 12 visits. All participants will use the patch at least once during the study. The drug efficacy will be evaluated by the percent change in pain intensity before and after treatment and by improvements in the following activities: daily life, walking, meal intake, mood regulation. The overall safety will be assessed based on the adverse events reporting.

ELIGIBILITY:
Inclusion Criteria:

* spine related and extremity pain lasting for 3 months or longer
* pain with Numeric Rating Scale (NRS) at 4 or higher in the past 72 hours
* good overall health condition based on the medical history and clinical laboratory tests
* participants using appropriate contraception in case of childbearing potential during the study period.

Exclusion Criteria:

* history of hypersensitive reaction to narcotic analgesics
* history of narcotic abuse
* serious psychotic disorder
* unable to use transdermal analgesics due to a dermatological condition
* history of CO2 retention (e.g., chronic obstructive pulmonary disease)
* surgery in the area with pain within 7 days prior to initiation of the clinical study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2005-10; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
The change in pain intensity | Baseline, 12 weeks
  The percent change in Pain Intensity Difference (PID) after study treatment (Week 12) compared to Day 0, prior to study treatment.

SECONDARY OUTCOMES:
Daily dose of prescribed medication | 12 weeks
  Change in daily dose of study medication prescribed at Day 0 and after 1, 4, 8 weeks.
Change in functionality | 12 weeks
  Satisfaction in functionality by participants evaluated at day 0 and after 1, 4, 8 and 12 weeks of treatment, measured as improvements in change of scores from 0 (not disturbing) to 10 (completely disturbing).
Change in sleep | 12 weeks
  Change in the frequency of waking up due to pain during the sleep.
Satisfaction in study medication | 12 weeks
  Satisfaction in study medication by participants and investigators summarized at Week 4, 8 and 12 visits.
The number of participants reporting adverse events (AEs) | 12 weeks
  All AEs during the study period will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd., Korea Clinical Trials, Study Director — Janssen Korea, Ltd., Korea
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Result] Park JH, Kim JH, Yun SC, Roh SW, Rhim SC, Kim CJ, Jeon SR. Evaluation of efficacy and safety of fentanyl transdermal patch (Durogesic D-TRANS) in chronic pain. Acta Neurochir (Wien). 2011 Jan;153(1):181-90. doi: 10.1007/s00701-010-0785-4. Epub 2010 Sep 7. PMID 20821238
- See also: Evaluation in Efficacy and Safety of Fentanyl-TTS (Durogesic® D-Trans) for Treatment of Chronic Pain — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=1148&filename=CR002155_CSR.pdf